CLINICAL TRIAL: NCT04174274
Title: Investigation of Compliance With Ventilator-Associated Pneumonia Prevention Methods and Incidence of Ventilator-Associated Pneumonia in Intensive Care Units
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Gokhan Erdem, residant, Diskapi Teaching and Research Hospital
Other Study IDs: VAP incidence and compliance
Record Dates: First submitted 2019-11-20; First posted 2019-11-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: The Incidence of Ventilator-associated Pneumonia and Rate of Compliance With Survey Criteria

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- positive: ventilator-associated pneumonia-developed group followed by mechanical ventilation
  Interventions: Other: ventilator-associated pneumonia-developed group followed by mechanical ventilation
- negative: not ventilator-associated pneumonia-developed group followed by mechanical ventilation
  Interventions: Other: not ventilator-associated pneumonia-developed group followed by mechanical ventilation

INTERVENTIONS:
Other: ventilator-associated pneumonia-developed group followed by mechanical ventilation — compliance with ventilator-associated pneumonia prevention methods and investigating the incidence of ventilator-associated pneumonia in intensive care units
  Groups: positive
Other: not ventilator-associated pneumonia-developed group followed by mechanical ventilation — compliance with ventilator-associated pneumonia prevention methods and investigating the incidence of ventilator-associated pneumonia in intensive care units
  Groups: negative

SUMMARY:
Ventilator-associated Pneumonia (VAP) is a high-mortality hospital infection that occurs in patients undergoing invasive Mechanical Ventilation (MV) and is frequently encountered in intensive care units. Prolonged mechanical ventilation, prolonged hospitalizations, excessive use of antibiotics and increased medical costs are seen. Therefore, compliance with ventilator-associated pneumonia prevention methods is becoming increasingly important. Therefore, in the investigator's study was to investigate compliance with ventilator-associated pneumonia prevention methods and the incidence of ventilator-associated pneumonia in intensive care units.

DETAILED DESCRIPTION:
In the first stage of the study, Diskapi Yildirim Beyazit Education and Research Hospital Anesthesia Reanimation 1-2-3-4, compliance with ventilator-associated pneumonia prevention rules in neurology, neurosurgery, and internal medicine intensive care units will be investigated. The researcher will visit the intensive care units included in the study twice a day (10:00 and 14:00) by Dr. Gökhan Erdem for 1 week at the same time of day and monitor whether they work in accordance with VAP prevention rules.

VAP prevention methods: Head angle 30-45 degrees, peptic ulcer prophylaxis, thromboembolism prophylaxis, daily wake up test, use of chlorhexidine in oral care, bacterial filter use in ventilator circuit, daily spontaneous breathing trials, silver-coated endotracheal tube use, cuff pressure adequacy, hand hygiene , VAP nurse training, avoiding excessive distension of the stomach, equipment contamination, mechanical tooth cleaning, daily assessment for patient separation from mechanical ventilation, sterile aspiration technique, use of sterile gloves before aspiration, aspiration of subglottic secretions will be recorded.

In the second stage of the study, Diskapi Yildirim Beyazit Education and Research Hospital anesthesia reanimation 1-2-3-4, demographic characteristics of all hospitalized patients for neurological, neurosurgery, and internal medicine intensive care units, reason for hospitalization in intensive care unit, APACHE score, duration of mechanical ventilation, length of stay in ICU unit, blood transfusion, urinary infection, wound infection, presence of infection in at least one site, duration and type of surgery if operated, post-op prophylactic antibiotic use, history of CPR, history of difficult intubation, shape and duration of intubation, presence of tracheostomy , time from intubation to tracheostomy opening, residence time in ICU, change of filters in mechanical ventilator circuits, antibiotic use, low serum albumin value, sedative use, steroid use, feeding type, inotropic requirement, prokinetic agent use, number of bed personnel and nurses, reentubation history, transport history, glaskow coma score, frequency of endotracheal aspiration, peep need, smoking history, nasogastric use, chest tube, central venous catheter, presence of arterial catheter, history of dialysis, continuous infusion therapy, aerosol therapy, chronic diseases will be recorded. Patients under 18 years of age who had previously been diagnosed with pneumonia, lung expansion devices such as cpap, nasal peep, hypocpap were not applied via tracheostomy or endotracheal intubation, and patients due to high frequency ventilation or extracorporeal life support were excluded from VAP surveillance.

ELIGIBILITY:
Inclusion Criteria:

* patients followed for more than 48 hours on a mechanical ventilator

Exclusion Criteria:

* previously diagnosed with pneumonia
* Patients under the age of 18
* Unless lung expansion devices such as cpap, nasal peep, hypo cpap are applied via tracheostomy or endotracheal intubation
* patients due to high frequency ventilation or extracorporeal life support

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients followed up on mechanical ventilation by tracheostomy or endotracheal intubation in ICUs aged 18 and over
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
Investigation of ventilator-associated pneumonia incidence in intensive care units | 01.12.2019-01.03.2020
  The development of ventilator-associated pneumonia leads to many negative conditions. Therefore, the incidence of ventilator-associated pneumonia is important in terms of decreasing hospital care costs, requiring longer mechanical ventilation, length of hospital stay, mortality and morbidity.

SECONDARY OUTCOMES:
Investigation of compliance with ventilator-associated pneumonia prevention methods in intensive care units | 01.12.2019-01.03.2020
  Compliance with ventilator-related pneumonia prevention rules will be investigated in the intensive care units of Diskapi Yildirim Beyazit Training and Research Hospital.

OTHER OUTCOMES:
Investigation of possible risk factors for ventilator-associated pneumonia | 01.12.2019-01.03.2020
  The parameters that may affect ventilator-associated pneumonia rates in patients who were supported by invasive mechanical ventilator in intensive care units of Diskapi Yildirim Beyazit Training and Research Hospital will be recorded.